CLINICAL TRIAL: NCT03663387
Title: PET Measures of CSF Clearance in Preclinical Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1804019181; 1RF1AG057570-01 (NIH)
Record Dates: First submitted 2018-08-10; First posted 2018-09-10 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood incl. geneting testing/APE Genotyping, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Normal subjects: 70

SUMMARY:
The purpose of this study is to measure cerebrospinal fluid (CSF) clearance. CSF cushions the brain from impact and carries waste products from the brain to the bloodstream. This process is known as clearance. Researchers have considered that impaired clearance of amyloid (a protein) from the aging brain causes buildup of amyloid in the brain and plays a role in increased risk for Alzheimer's disease. However, until recently, there has not been a method to measure CSF clearance. This study will examine CSF clearance using positron emission tomography (PET) scanning, which creates images of structures in the body and their functioning. This study will also measure the amount of two proteins, tau and amyloid, in the brain. Tau and amyloid are proteins that build up in the brains of people with Alzheimer's disease. An investigational compound (tracer) called [18F]MK-6240 is injected into the blood prior to the scan in order to take images of the CSF clearance and measure tau protein in the brain. This tracer is considered investigational because it is not approved by the US Food and Drug Administration (FDA) for clinical use and is only being used for research purposes.

DETAILED DESCRIPTION:
The impaired clearance of amyloid-β (Aβ) leading to the accumulation of Aβ plaques and consequent neurodegeneration, is a partially understood mechanistic hypothesis for late onset Alzheimer's disease (AD). Using Positron Emission Tomography (PET) and a tracer for tau lesions, with a low molecular weight that rapidly enters and clears the brain, the investigators developed, replicated, and validated a non-invasive method to estimate the clearance of CSF at ventricular and brain levels. The investigators propose to complete over five years, a 2y longitudinal study designed to test in preclinical AD the hypothesis that reduced CSF clearance measured with the tau tracer [18F]-MK6240 is predictive of: a) future amyloid lesions (PiB-PET or Florbetaben-PET); b) brain atrophy (MRI); and c) cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 20-100 years old will be enrolled. Younger subjects are not included as the risk for brain amyloid lesions is too low
* All subjects will speak English as their first language or demonstrate proficiency in English.
* All subjects may have normal cognition or cognitive impairment.
* All subjects will be in good general health and able to participate in the LP and imaging exams. This determination is made by the study neurologist and reviewed at a consensus meeting for each subject.

Exclusion Criteria:

* Uncontrolled hypertension or metabolic disease
* Neurodegenerative disorders (i.e. Parkinson disease. LBD, or FTD).
* Long life major depression. Baseline scores ≥20 on Beck Depression Inventory at baseline
* Long-life DSM-IV axis 1 disorders.
* Mental retardation.
* Substance abuse.
* Concurrent medication limiting validity of neuropsychological tests or imaging.
* Anti-depressants with anti-cholinergic properties
* Monoamine oxidase inhibitors (MAOi)
* Regular use of narcotic analgesics (>2 doses per week).
* Use of neuroleptics
* Individuals taking over the counter memory enhancing or protecting medications (e.g. ginkgo biloba, vitamins) are not excluded.
* Implanted medical devices that are incompatible with MRI imaging.
* Radiation exposures exceeding annual Rad Worker limits.
* Heart failure stage D as defined by American Heart Association (7).
* Chronic kidney disease in stages ≥ 4, as defined per National Kidney Foundation (8).
* Brain tumor and other neoplastic disorders outside the brain where disease itself or its treatment (radiation, chemotherapy) is likely to affect brain structure or function.
* Stroke when meeting criteria for total anterior, partial anterior or posterior circulation infarct according to the Oxford Community Stroke Project classification. Patients with clinically silent of lacunar strokes and transient ischemic attacks will not be excluded.
* Significant head trauma.
* Hydrocephalus.
* Hostility or refusal to cooperate
* Person's receiving chronic anti-coagulation therapy
* Person's participating in other research projects will be excluded when the other project(s) 1) involve radiation exposure which in combination with the current project would increase radiation exposure above federal guidelines, 2) involve administration of study drug or other experimental therapy, or 3) prohibit participation in other research projects.
* Participants in this study will be allowed to participate in other observational research studies. The investigators will review at enrollment the full array of projects a subject may be involved in and inform the other PI's to ensure that subject safety and research data integrity is not compromised.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve male and female volunteer subjects from any racial or ethnic group with a diagnosis normal cognition or mild cognitive impairment. The proposed sample is not intended to be representative of a general population, but it will approximate the samples recruited in NIH and industry sponsored FDA approved clinical trials targeting secondary AD prevention. At this stage of knowledge of human brain CSF clearance, a population based approach was considered premature and over cap funding to support a larger study was not permitted for RFA AG-17-055. Rather, our design uses Aβ enrichment to enable an efficient test of the CSF clearance hypothesis in a clinically relevant group.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Percent change in brain amyloid | Baseline and 24 Months follow-up
  Percent change in brain amyloid measured by positron emission tomography
Percent change in cortical ribbon thickness | Baseline and 24 Months follow-up
  Percent change in cortical ribbon thickness measured by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Mony J de Leon, ED.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available through the Brain Health Imaging Institute at Weill Cornell Medicine through correspondence with mdl4001@med.cornell.edu
Access Criteria: Anyone who wishes to access the data who will provide a methodologically sound proposal.